CLINICAL TRIAL: NCT07190872
Title: Sleep Hygiene Among Undergraduate Students Studying in the Health Field: A Study on Awareness and Behavioural Change
Brief Title: Sleep Hygiene in Undergraduate Students Studying in the Field of Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Dilek Gümüş, Assistant professor, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BilecikSeyhEU-CH-DG-01
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Sleep Hygiene
Keywords: sleep hygiene; sleep quality; behavior change; transtheoretical model
MeSH Terms: conditions — Sleep Hygiene; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study has a single-arm, pre-post design (allocation: N/A, masking: none). Participants will be selected from among volunteer students in the 2nd-year day programs of the SHMYO. All participants receive two sessions of in-class training (each ~40 minutes; total 80 minutes). The intervention consists of the following components: providing information, increasing awareness, creating an individual sleep plan, and supporting maintenance with short assignments, all within the framework of the Transtheoretical Model. Assessments are performed at T0 (baseline), T1 (2 weeks), and T2 (4 weeks). Primary outcomes: Change in Sleep Hygiene Index and PSQI scores; secondary outcomes: Relationships with Sleep Hygiene Information Test score and lifestyle variables (caffeine, screen time, perceived stress). The analysis is conducted using within-participant comparisons (e.g., paired tests/repeated measures). The aim is to demonstrate the effect of a brief, structured educational model on sleep hygie
Who Masked: Outcomes Assessor
Masking Description: Since this study is a single-arm design based on an educational intervention, blinding is not applied to participants or researchers. All students participate in the same training session and fill in their own data. However, during the statistical analysis phase, an independent expert outside of the researcher will work on de-identified (anonymous) data. Thus, the participants' identities will be kept confidential, and the evaluation will be based solely on coded data. No individual names or identifying information will be included in the research reports.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Hygiene Education (Experimental Intervention Arm) (Experimental): Students in the intervention group will receive face-to-face sleep hygiene education in a total of 4 sessions, once a week for 40 minutes over a period of four weeks. The education is designed within the framework of the Transtheoretical Model and focuses on topics such as the concept of sleep hygiene, regular sleep hours, limiting caffeine and screen use, organizing the sleep environment, and stress management. The training will be provided by a nurse experienced in sleep health.
  Interventions: Behavioral: sleep hygiene education
- Control Group (No Intervention): Students in the control group will not receive any educational intervention or message support during the study period; they will continue with their daily routines. Assessments are conducted at the same time points as the intervention group. After the study is completed, the same training materials will be made available to the control group.

INTERVENTIONS:
Behavioral: sleep hygiene education — Students in the intervention group will receive face-to-face sleep hygiene training in a total of 4 sessions, once a week for 40 minutes over a period of four weeks. The education is designed within the framework of the Transtheoretical Model and focuses on topics such as the concept of sleep hygiene, regular sleep hours, limiting caffeine and screen use, organizing the sleep environment, and stress management. The training will be provided by a nurse experienced in sleep health.
  Arms: Sleep Hygiene Education (Experimental Intervention Arm)

SUMMARY:
This study looks at sleep hygiene-the daily habits and environment that help people sleep well-among 2nd-year students at the Health Services Vocational School of Bilecik Şeyh Edebali University (Türkiye). Many health sciences students have busy schedules, clinical practice, and exam stress, which may reduce sleep quality. Good sleep is important for learning, attention, mood, and overall health.

Purpose:

The aim is to assess the current sleep hygiene and quality of students, and determine whether a brief, in-person education program can enhance their knowledge, habits, and sleep quality in the upcoming weeks.

Who can take part:

The program is designed for daytime (normal education) 2nd-year students in programs such as Operating Room Services, Paramedic, Opticianry, Pharmacy Services, Medical Laboratory Techniques, Medical Documentation and Secretariat, and Child Development who volunteer and give written consent. Participation is voluntary, and you may leave the study at any time without any penalty.

What will happen if you join:

You will complete short forms before the education session to measure sleep habits and sleep quality (for example, bedtime, caffeine use, and screen time).

You will attend four classroom sessions (each about 40 minutes). These sessions explain practical sleep tips (regular bed/wake times, reducing evening caffeine and screen time, preparing a quiet/dark room, simple relaxation after clinical shifts) and help you create a personal sleep plan.

You will fill out the same forms again 2 weeks and 4 weeks after the education to see changes over time.

What we measure:

Sleep hygiene behaviors (how often helpful/unhelpful habits are used)

Sleep quality refers to how restful sleep feels, the time it takes to fall asleep, the frequency of night awakenings, and overall daytime functioning.

Knowledge about sleep hygiene (a short quiz) We will also look at factors like stress level, evening screen use, and caffeine intake.

Possible benefits:

You may learn practical ways to improve sleep, which can help with attention, mood, and daily performance.

Possible risks/discomforts:

This is an educational program. Risks are minimal (for example, brief discomfort when answering personal questions about sleep). You can skip any question you do not want to answer.

Privacy:

All information will be kept confidential and used only for research. Reports will not include names or identifying details.

Costs and payment:

There is no cost to taking part, and there is no payment for participation.

Withdrawal:

Participation is voluntary. You may stop at any time without affecting your courses or grades.

DETAILED DESCRIPTION:
Sleep Hygiene in Associate Degree Students in the Health Field: A Study on Awareness and Behavioral Change Introduction Sleep is an integral part of human life, serving as a fundamental requirement for physical health, mental acuity, and emotional balance. Sufficient and quality sleep offers a wide range of positive effects, from strengthening the immune system to supporting cognitive functions, while sleep deprivation or disorders seriously threaten individuals' daily lives (Walker, 2017). Factors such as technological dependence brought about by modern life, intense work pace, and stress negatively affect sleep hygiene, especially in young adults. Research conducted in Turkey shows that the sleep quality of the young population is low, and this is associated with mental health problems such as stress, anxiety, and depression (Ağargün et al., 1996; Özdemir et al., 2015). These findings are also supported in the current literature; for example, Kaya and Bozkurt (2021) revealed the prevalence of sleep problems among university students in Turkey and its connection to academic performance. This situation highlights the critical importance of sleep hygiene, especially for groups facing both academic and professional pressures, such as associate degree students.

Students at the Health Services Vocational School (SHMYO) have a demanding schedule with additional responsibilities such as practical training and internships, alongside theoretical courses. These students need skills such as attention, concentration, and emotional resilience due to their future professions; however, the long hours of internships, exam stress, and irregular daily routines disrupt their sleep patterns, putting these skills at risk. A recent study reported that the sleep quality of students studying in the healthcare field is lower compared to the general university population, and this is associated with occupational burnout (Al-Maddah et al., 2022). Additionally, Kaya and colleagues (2023) reported that over 60% of healthcare students in Turkey sleep less than the recommended 7-9 hours, which reduces their ability to cope with stress. Sleep hygiene, in this context, is defined as the behaviors and environmental adjustments individuals develop to optimize their sleep quality (Mastin et al., 2006). While there is evidence in the literature that sleep hygiene education increases awareness and improves sleep quality (Brown et al., 2006; Irish et al., 2020), the impact of such interventions on associate degree students studying in the healthcare field in Turkey has not been adequately researched.

This deficiency highlights a significant literature gap in understanding the impact of sleep hygiene on students and developing effective educational strategies. Although international studies have shown that sleep hygiene education improves sleep habits and increases academic performance in university students (Hershner and Chervin, 2020), such studies in Turkey have generally focused on the general university population, neglecting specific groups like health students. For example, Özcan and Kaya (2022) reported that sleep hygiene was inadequate among university students in Turkey and worsened after the pandemic; however, no analysis specific to health students was presented. This study aims to fill this gap by targeting second-year students in the regular education program at Bilecik Şeyh Edebali University's Vocational School of Health Services. Considering the importance of sleep hygiene for the professional success and personal health of health students, raising awareness and changing behavior in this group can benefit both individuals and society.

This study was designed within the framework of the Transtheoretical Model (Prochaska and DiClemente, 1983). The model systematically addresses the stages individuals go through in the process of behavior change (awareness, preparation, action, maintenance) and offers an effective way to develop habits such as sleep hygiene. In this context, the aim is to increase students' awareness of sleep hygiene, assess their current habits, and examine the effects on long-term behavioral changes by implementing a multi-session face-to-face training program. The study will adhere to ethical guidelines, be based on the principle of voluntary participation, and protect the confidentiality of participants, and the data will be used solely for scientific purposes. In this direction, it is aimed to develop comprehensive educational strategies for acquiring healthy sleep habits by analyzing the changes that will occur in students' knowledge, attitudes, and behaviors regarding sleep hygiene. Thus, while supporting the academic success and professional competence of health students, a unique contribution will be made to the literature on sleep hygiene awareness in Turkey.

Method This study was designed to assess the sleep hygiene awareness of 2nd-year students studying in regular education programs at Bilecik Şeyh Edebali University Health Services Vocational School and to examine the effect of a multi-session face-to-face training on this awareness. The research was conducted using a quantitative method and an experimental design.

Research Purpose The purpose of this study is to determine the current sleep hygiene awareness among second-year students in the Health Services Vocational School's regular education program, to examine students' sleep habits and knowledge levels, and to reveal the long-term effects of multi-session face-to-face education on this awareness and behavioral change. In this way, it is aimed to develop comprehensive educational strategies for acquiring healthy sleep habits by evaluating the positive changes in students' knowledge, attitudes, and behaviors regarding sleep hygiene.

Research Questions What are the current levels of sleep hygiene awareness among students? How does the multi-session face-to-face training application affect students' level of awareness and behaviors regarding sleep hygiene? Are statistically significant and lasting changes observed in students' knowledge, attitudes, and behaviors related to sleep hygiene after the training? Is there a relationship between students' knowledge levels of sleep hygiene and their daily sleep habits? Through which factors (e.g., stress, caffeine consumption) does the impact of education become more pronounced? Research Universe and Sample The research universe consists of 2nd-year students enrolled in regular education programs at Bilecik Şeyh Edebali University Health Services Vocational School (SHMYO). In this context, the programs within the SHMYO (Operating Room Services, First and Emergency Aid, Opticianry, Pharmacy Services, Medical Laboratory Techniques, Medical Documentation and Secretarial, and Child Development) have been targeted. The sample will be determined by a random selection method from students who are accessible during the study period and volunteer to participate in the research. The sample size will be calculated using power analysis to ensure the reliability of the statistical analyses; a medium effect size (Cohen's d = 0.5) and a power assumption of 80% will be targeted, with a minimum of 50 students. Diversity will be ensured by representative participation from different programs.

Data Collection Tools and Data Collection Data will be collected using the "Student Life and Sleep Factors Form," the "Sleep Hygiene Index (SHI)," the "Pittsburgh Sleep Quality Index (PSQI)," and the "Sleep Hygiene Knowledge Test." Student Life and Sleep Factors Form: Developed by researchers through a literature review, it was prepared to assess basic demographic and social information relevant to the study's aims and questions. The form includes information such as participants' age, gender, height, weight, program of study (e.g., Medical Laboratory Techniques), chronic health problems, regular medication use, place of residence, whether they have previously received training on sleep hygiene, daily caffeine consumption (☐ None ☐ 1-2 cups ☐ 3-4 cups ☐ 5 or more), screen use in the last 2 hours before bed (☐ No ☐ Yes, <30 min ☐ Yes, 30-60 min ☐ Yes, >60 min), weekly class/study hours (____ hours), and stress level in the last month (☐ Very low ☐ Low ☐ Medium ☐ High ☐ Very high). These questions, covering the fundamental variables that affect sleep hygiene and quality, enable the assessment of the roles of caffeine (Mastin et al., 2006), screen time (Walker, 2017), and academic load and stress (Özdemir et al., 2015), providing data for the analysis of the impact of education and the knowledge-behavior relationship (Buysse et al., 1989).

Sleep Hygiene Index (SHI): Developed by Mastin et al. (2006), the Turkish validity and reliability study was conducted by Özdemir et al. (2015). The scale, consisting of 13 items evaluated using a five-point Likert scale, measures how frequently participants engage in behaviors related to sleep hygiene. The scores obtained range from 13 to 65, with higher scores indicating poorer sleep hygiene. The scale is derived from the diagnostic criteria for inadequate sleep hygiene found in the International Classification of Sleep Disorders. The Cronbach's alpha coefficient was calculated as 0.70, indicating a valid and reliable scale (Özdemir, Boysan, and Güleç, 2015).

Pittsburgh Sleep Quality Index (PSQI): Developed by Buysse et al. (1989), the Turkish validity and reliability study was conducted by Ağargün et al. (1996). The scale was developed to assess individuals' sleep quality and potential sleep disorders and consists of 19 self-report items and 7 components. These components are listed as subjective sleep quality, sleep latency (time to fall asleep), sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication use, and daytime dysfunction. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality. The Cronbach's alpha coefficient was calculated as 0.80, indicating a valid and reliable scale (Ağargün, Kara, and Anlar).

Sleep Hygiene Knowledge Test: This test, developed by researchers, is a 10-item test that measures basic knowledge about sleep hygiene (e.g., the effects of caffeine and screen time). This test was added to directly assess the level of knowledge.

The data collection process will be carried out using the pre-test-post-test method; the pre-test will be administered before the training, and the post-tests will be administered 2 weeks and 4 weeks after the training. As part of the intervention, a multi-session training program detailed below will be conducted, and brochures will be distributed.

Educational Intervention The educational intervention aims to increase students' awareness of sleep hygiene and behavioral changes. It will be delivered face-to-face in two sessions (40 minutes each, 80 minutes total) for the target audience. The content, designed based on the Transtheoretical Model, was developed using UHI and PSQI data, supported by literature, and adapted to students' living conditions (e.g., practical course load).

ELIGIBILITY:
Inclusion Criteria:

* Being an associate degree student at Bilecik Şeyh Edebali University School of Health Services.

Being a student who has started clinical practice and is actively doing an internship in the clinic.

Being between the ages of 18 and 25

Scoring ≥ 30 on the Sleep Hygiene Index (UHI) (poor sleep hygiene score)

Agreeing to volunteer for the study and signing the informed consent form

Not having received any sleep hygiene training in the last 3 months.

Being able to participate regularly in the research process (pre-test, training intervention, and post-tests).

Exclusion Criteria:

* Having been diagnosed with a sleep disorder (e.g., insomnia, sleep apnea, narcolepsy, etc.).

Receiving a diagnosis of a psychiatric illness that can affect mental health and/or taking psychiatric medication regularly.

Having a chronic illness and taking regular medication (e.g., diabetes, epilepsy, cardiovascular diseases).

Working nite shifts or having irregular sleep schedules (e.g., students on duty).

Declaring that they will be unable to regularly participate in the study process or failing to comply with interventions during the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Total score on the Sleep Hygiene Index | Baseline (T0) → Week 4 (T2). Interim analysis: Week 2 (T1); optional long-term: Month 3 (T3). The primary analysis is on T2.
  The Sleep Hygiene Index is a 13-item, 5-point Likert scale; the total score is 13-65, with a higher score indicating poorer sleep hygiene. Turkish validity and reliability have been reported. The primary outcome is the within-participant total UHI score change (T2-T0) and the between-group mean change difference (intervention - control; negative values indicate improvement). The scale is administered in the classroom setting using standard instructions and in self-report format.

IPD SHARING:
Plan to Share IPD: No